CLINICAL TRIAL: NCT02191046
Title: A Randomized- Controlled Study Comparing the Effect of Squeezable Bottle Nasal Irrigation Device With Syringe in Children With Sinusitis
Brief Title: Effect of Squeezable Bottle Nasal Irrigation Device in Children With Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, araya satdhabudha, clinical professor, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ทป 45/2555; 45/2555 (Other Grant/Funding Number: Thammasat research grant)
Record Dates: First submitted 2014-07-13; First posted 2014-07-15 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Sinusitis
Keywords: nasal irrigation; sinusitis; children; buffered hypertonic saline; nasal irrigation device
MeSH Terms: conditions — Sinusitis | interventions — Syringes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- syringe 20 ml (Active Comparator): nasal irrigation with syringe by using buffer hypertonic saline about 100-240 ml until no nasal discharge
  Interventions: Device: syringe 20 ml
- squeezable bottle (Experimental): nasal irrigation with squeezable bottle by using buffer hypertonic saline about 100-240 ml until no nasal discharge
  Interventions: Device: squeezable bottle

INTERVENTIONS:
Device: squeezable bottle — nasal irrigation twice daily for 2 weeks period
  Other Names: EEZNIS
  Arms: squeezable bottle
Device: syringe 20 ml — nasal irrigation twice daily for 2 weeks
  Arms: syringe 20 ml

SUMMARY:
The purpose of this study is to the effect of squeezable bottle nasal irrigation device with syringe in children with sinusitis in symptom score and satisfaction to nasal irrigation

DETAILED DESCRIPTION:
sinusitis is the one of common diseases in Thailand. Nasal irrigation has been used as an adjunctive treatment.In previous study shown that buffer hypertonic nasal irrigation have more effective to decrease symptom in patient sinonasal disease when compare to normal saline.Until now, there are no clear data comparing the effectiveness on sinonasal symptom of the various devices use in children with sinusitis. The purpose of this study was to compare the effect of squeezable bottle nasal irrigation device with syringe in children with sinusitis in symptom score and satisfaction to nasal irrigation.

ELIGIBILITY:
Inclusion Criteria:

1. age 3-15 years
2. diagnose sinusitis by each of following criteria 2.1 persistent upper respiratory infection symptoms > or = 10 days 2.2. severe upper respiratory infection symptom with greenish discharge per nose or periorbital swelling 2.3 double sickening of upper respiratory infection symptoms

Exclusion Criteria:

1. patient who has history of penicillin allergy
2. patient who has complication of sinusitis
3. patient with a history of nasal anatomical defects
4. patient who has immune deficiency or primary ciliary dyskinesia

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Araya Satdhabudha, MD, Principal Investigator — Thammasat University
Locations (1):
- Araya Satdhabudha, Klongluang, Pratumthanee, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: we enrolled sinusitis patient age 3-15 year during March 2013 - May 2014. We excluded patients with a history of penicillin allergy, nasal anatomic defects, immunodeficiency or had complication from sinusitis. Patient with low compliance defined as the rate usage nasal irrigation estimated at less than 80% were excluded
Groups:
- Syringe 20 ml: nasal irrigation with syringe by using buffer hypertonic saline about 100-240 ml until no nasal discharge
  syringe 20 ml: nasal irrigation twice daily for 2 weeks period
Period: Overall Study
Arm/Group | Syringe 20 ml | Squeezable Bottle
Started | 41 | 39
Completed | 36 (exclude 5 patients because low compliance) | 38 (exclude 1 patient because low compliance)
Not Completed | 5 | 1
Not completed — low compliance | 5 | 1

BASELINE CHARACTERISTICS:
Population: Eighty sinusitis children participated in the study. 74 participants were finally assessed. six participants were discontinue irrigated their nose during treatment due to the nasal symptoms score improve; one patient from squeezable bottle group, five patients from disposable syringe group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Syringe 20 ml | Squeezable Bottle | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 38 | 74
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 25 | 22 | 47
Region of Enrollment [Number; unit: participants]
  Thailand | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: the Effect of Squeezable Bottle and Syringe on Clinical Effectiveness in Sinusitis Children
Description: For 5S-score, we measured the the mean 5-s score of both group at 2 weeks compare to the mean 5-s score at baseline visit and compare 5S-score between group at 2 weeks. The S5- score is a scale assessing severity of sinusitis. It compose of the symptom scores for nasal obstruction, day and nighttime cough, headache and nasal discharge. All symptom were graded from 0(no symptom) to 3 (severe ).The score were summed to give the mean 5S-score.It range from 0 (best possible outcome) to 15(worst possible outcome). 7-point Likert scale for satisfaction score is scale from 1 (indicating unsatisfactory) to 7 (indicating excellent). For satisfaction, we reported the result in the term of 7 points Likert scale and compare these scale between group at 2 weeks after treatment
Time Frame: compare 5S-score of both group at 2 week and at baseline visit .compare the mean 5S-score and satisfaction score between both group at 2 weeks after treatment
Population: The S5- score is the symptom scores for nasal obstruction, day and nighttime cough, headache and nasal discharge. All symptom were graded from 0(no symptom) to 3 (severe ).The score were summed to give the mean 5S-score.7-point Likert scale for satisfaction score is scale from 1 (indicating unsatisfactory) to 7 (indicating excellent).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Syringe 20 ml: improve 5-s score at 2 week period after treatment when compare to the beginning status with minimal side effect
- Squeezable Bottle: improve 5-s score at 2 week period after treatment when compare to the beginning status with minimal side effect and significant improve in 5-s score and satisfaction when compare to syringe group
Arm/Group | Syringe 20 ml | Squeezable Bottle
Number analyzed (Participants) | 36 | 38
units on a scale
  5S-score at baseline | 6.56 (2.35) | 6.89 (2.49)
  5S-score at 2 weeks | 2.17 (2.03) | 1.24 (1.55)
  satisfaction score at baseline | 5.11 (1.19) | 5.97 (1.31)
  satisfaction score at 2 weeks | 6.11 (0.85) | 6.57 (0.64)
Statistical Analysis 1: Comparison: Syringe 20 ml; compare the mean 5S-score between before and after treatment in syringe group; Test type: Non-Inferiority or Equivalence — power of study = 90%; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 4.38, 95% CI 2-sided [3.41 to 5.37], Standard Deviation 2.89
Statistical Analysis 2: Comparison: Syringe 20 ml vs Squeezable Bottle; compare the mean 5S-score between 2 groups at 2 weeks after treatment; Test type: Non-Inferiority or Equivalence — power of study = 90%; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.93, 95% CI 2-sided [0.094 to 1.76], Standard Deviation 0.42
Statistical Analysis 3: Comparison: Syringe 20 ml vs Squeezable Bottle; satisfaction score between two groups at 2 weeks after treatment; Test type: Non-Inferiority or Equivalence — power of study = 90%; p < 0.05, t-test, 2 sided; Mean Difference (Net) = -0.47, 95% CI 2-sided [-0.82 to -0.12], Standard Deviation 0.17
Statistical Analysis 4: Comparison: Squeezable Bottle; compare the mean 5s-score between before and after treatment in squeezable bottle group; Test type: Non-Inferiority or Equivalence — power fo study = 90%; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 5.66, 95% CI 2-sided [4.62 to 6.69], Standard Deviation 3.16

2. Secondary Outcome: the Contamination in Nasal Irrigation Devices
Description: compare the result of bacterial culture in both group of nasal irrigation devices. We reported in the following item; no growth, gram positive or gram negative or mixed organism
Time Frame: at second week after treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: we monitor side effect from the beginning of treatment until 2 weeks after treatment
Description: we monitor side effect from the beginning of treatment until 2 weeks after treatment. the physician asking the symptoms after nasal irrigation at baseline visit then the symptoms were recorded daily by parents and noted in diary card
Groups:
- Syringe 20 ml; Squeezable Bottle: record adverse event at baseline and daily adverse events until 2 weeks after treatment
Arm/Group | Syringe 20 ml | Squeezable Bottle
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 8/36 | 7/38
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Syringe 20 ml (N=36) | Squeezable Bottle (N=38)
nasal irritation (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 2 (3)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (5)
tinnitus (Ear and labyrinth disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes